CLINICAL TRIAL: NCT06538311
Title: Neuromodulation of Brain Function in Alzheimer's Disease and Related Dementias
Brief Title: Transcranial Magnetic Stimulation Treatment for Alzheimer's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alexandra Touroutoglou, Assistant Professor of Neurology, Harvard Medical School (HMS and HSDM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022A002983
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Logopenic Progressive Aphasia; Amnestic Symptoms
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Within-subject crossover design
Masking Description: Through use of SHAM rTMS stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- AD, aMCI, lvPPA patients, and preclinical AD (Experimental): All participants will receive the same study interventions in a within-subject crossover design.
  Interventions: Device: Active rTMS; Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS — All study participants will receive one block of ACTIVE rTMS. Each block will consist of daily sessions of active rTMS delivered to the left dorsolateral prefrontal cortex over ten days (Monday through Friday).
Device: Sham rTMS — All study participants will receive one block of SHAM rTMS. Each block will consist of daily sessions of SHAM rTMS delivered to the left dorsolateral prefrontal cortex over ten days (Monday through Friday).

SUMMARY:
In this research study we want to learn more about the effects of non-invasive brain stimulation on memory and brain-network function in cognitively unimpaired older adults and in patients with amnestic mild cognitive impairment (aMCI).

This study will use a form of non-invasive brain stimulation called repetitive Transcranial Magnetic Stimulation (rTMS). rTMS will slightly alter activity in an area of your brain that controls memory. Changes resulting from this stimulation will be measured with behavioral tests of memory and general cognition, as well as by taking images of your brain with Magnetic Resonance Imaging (MRI).

Participants will come in for one baseline visit followed by 10 days of daily rTMS study visits (Monday through Friday) and an evaluation visit. Then, there will be a 2-week break. After this break, they will return for another baseline visit, an additional 10 days of rTMS, and a final evaluation visit.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 40-99
2. Native English speakers
3. Willing and able to consent to the protocol and undergo imaging and neuropsychological testing at the specified time points
4. Patients with PPA will be asked to bring a study partner to all visits
5. Patients with very mild or mild PPA, patients with amnestic mild cognitive impairment and cognitively unimpaired participants with preclinical AD will be included.

Exclusion Criteria:

1. History of head trauma involving loss of consciousness or alteration in consciousness
2. Another major neurologic or psychiatric condition
3. Known presence of a structural brain lesion (e.g. tumor, cortical infarct)
4. Any contraindication to MRI, such as presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments, or foreign objects in the eyes, skin, or body
5. Longstanding premorbid history (i.e. longer than 10 years) of alcohol or substance abuse with continuous abuse up to and including the time that the symptoms leading to clinical presentation developed
6. Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the study protocol.
7. Unwilling to return for follow-up, undergo neuropsychological testing, TMS, and MR imaging
8. History of unprovoked seizures (i.e., seizures that occur in the absence of a clear provocation such as hyponatremia, hypoglycemia, etc.).
9. Subjects who have a first degree relative (e.g., father, mother or sibling) with a seizure disorder.
10. Subjects currently taking, or plan to take, medications which are highly epileptogenic. These include: clozapine, high doses of bupropion (i.e., greater than 400mg daily), diphenhydramine, cyclosporine, isoniazid, imipenem, chloroquine, tramadol and theophylline.
11. Subjects actively on anti-amyloid treatments. This is because they are at risk for bleeding due to amyloid-related imaging abnormalities (ARIA) that could provoke seizures.

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Memory | Baseline and post-treatment Day 11
  This will include observed changes in memory as a result of the stimulation through neuropsychological testing.
Changes in Brain Network Connectivity | Baseline and post-treatment Day 11
  This will include observed changes in resting-state functional connectivity as a result of the stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang JX, Rogers LM, Gross EZ, Ryals AJ, Dokucu ME, Brandstatt KL, Hermiller MS, Voss JL. Targeted enhancement of cortical-hippocampal brain networks and associative memory. Science. 2014 Aug 29;345(6200):1054-7. doi: 10.1126/science.1252900. PMID 25170153
- [Background] Damoiseaux JS, Prater KE, Miller BL, Greicius MD. Functional connectivity tracks clinical deterioration in Alzheimer's disease. Neurobiol Aging. 2012 Apr;33(4):828.e19-30. doi: 10.1016/j.neurobiolaging.2011.06.024. Epub 2011 Aug 16. PMID 21840627